CLINICAL TRIAL: NCT01153971
Title: An Open-label Study of Fludarabine and Cyclophosphamide Plus MabThera Followed by Maintenance With MabThera on Failure-free Survival in Treatment-naïve Patients With Advanced Indolent B-cell Nonfollicular Lymphoma
Brief Title: A Study of Induction and Maintenance Treatment With MabThera (Rituximab) in Patients With Indolent B-Cell Nonfollicular Lymphomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18324
Record Dates: First submitted 2010-06-14; First posted 2010-06-30 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-06

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: rituximab

INTERVENTIONS:
Drug: rituximab — 1
  Other Names: MabThera/Rituxan

SUMMARY:
This study will evaluate the efficacy and safety of MabThera in combination chemotherapy, followed by maintenance treatment with MabThera. The anticipated time on study treatment is 1-2 years, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients 18-65 years of age;
* previously untreated indolent nonfollicular non-Hodgkin's lymphoma;
* active disease;
* >=3 involved sites.

Exclusion Criteria:

* typical chronic lymphocytic leukemia;
* other malignancies within 3 years before study, except basal or squamous cell skin cancer or cancer in situ of the cervix;
* systemic corticosteroid use for >1 month;
* significant cardiovascular disease;
* central nervous system involvement;
* hepatitis B or C virus infection, or HIV infection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2005-07-20 (Actual); Primary Completion 2010-09-24 (Actual); Study Completion 2010-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (15):
- Italy (15):
  - Ospedale Civile Dello Spirito Santo; Divisione Di Ematologia, Pescara, Abruzzo
  - Ospedale Civile; Divisione Di Oncologia, Pescara, Abruzzo
  - Ospedale Oncologico Regionale; U.O. Oncologia Medica Ed Ematologia, Rionero in Vulture, Basilicate
  - Ospedale Riuniti; Divisione Di Ematologia, Reggio Calabria, Calabria
  - A.O.U. Policlinico di Modena-Dipartimento di Medicina Diagnostica, Clinica e di Sanità pubblica, Modena, Emilia-Romagna
  - Az. Osp. Arcispedale S. Maria Nuova; U.O. Di Ematologia, Reggio Emilia, Emilia-Romagna
  - Universita' Degli Studi La Sapienza-Ist.Di Ematologia;Dip. Biotecnologie Cel CELLULARI ED EMATOLOGIA, Rome, Lazio
  - A.O. Spedali Civili Di Brescia-P.O. Spedali Civili;U.O. Ematologia, Brescia, Lombardy
  - Ospedale Maggiore Di Milano; U.O. Ematologia I - Padiglione Marcora, Milan, Lombardy
  - Asst Grande Ospedale Metropolitano Niguarda; Dipartimento Di Ematologia Ed Oncologia, Milan, Lombardy
  - Ospedale Civile SS. Antonio E Biagio DI Alessandria; Ematologia, Alessandria, Piedmont
  - Az. Osp. S. Croce Ospedale Generale; Sezione Di Ematologia, Cuneo, Piedmont
  - A.O. Universitaria S. Giovanni Battista-Molinette Di Torino; Ematologia 1, Turin, Piedmont
  - Az. Osp. Papardo; Struttura Complessa Di Ematologia, Messina, Sicily
  - Az. Osp. Di Careggi; Divisione Di Ematologia, Florence, Tuscany

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab + Fludarabine + Cyclophosphamide: Cycle 1 (28-day cycle): Participants received fludarabine 25 milligrams per square meter (mg/m^2) intravenously (IV) and cyclophosphamide 250 mg/m^2 IV on Days 1, 2, and 3 and rituximab 375 mg/m^2 IV on Day 8, followed by 20 days of rest. Cycles 2-3 and Cycle 6 (28-day cycle): Participants received rituximab 375 mg/m^2 IV on Day 1 and fludarabine 25 mg/m^2 IV and cyclophosphamide 250 mg/m^2 IV on Days 2, 3, and 4 followed by 24 days of rest. Cycles 4-5 (28-day cycle): Participants received fludarabine 25 mg/m^2 IV and cyclophosphamide 250 mg/m^2 IV on Days 2, 3, and 4 and rituximab 375 mg/m^2 IV on Day 14, followed by 14 days of rest. Cycles 7-10 (2-month cycle): Following 2 months rest after the completion of Cycle 6, participants with complete response (CR), unconfirmed complete response (CRu), or partial response (PR), received maintenance therapy with rituximab 375 mg/m^2 IV on Day 1, followed by 2 months rest; cycle was repeated 4 times.
Period: Induction Phase (Months 1 to 7 of Study)
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Started | 47
Completed | 44
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1
Period: Maintenance Phase (Months 8-16 of Study)
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Started | 44
Completed | 41
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Clinical relapse | 1
Period: Follow-up (Months 17-40 of Study)
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Started | 41
Completed | 37
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 1
Not completed — Disease progression | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population: all enrolled participants who completed at least 2 cycles of treatment.
Groups:
- Rituximab + Fludarabine + Cyclophosphamide: Cycle 1 (28-day cycle): Participants received fludarabine 25 mg/m^2 IV and cyclophosphamide 250 mg/m^2 IV on Days 1, 2, and 3 and rituximab 375 mg/m^2 IV on Day 8, followed by 20 days of rest. Cycles 2-3 and Cycle 6 (28-day cycle): Participants received rituximab 375 mg/m^2 IV on Day 1 and fludarabine 25 mg/m^2 IV and cyclophosphamide 250 mg/m^2 IV on Days 2, 3, and 4 followed by 24 days of rest. Cycles 4-5 (28-day cycle): Participants received fludarabine 25 mg/m^2 IV and cyclophosphamide 250 mg/m^2 IV on Days 2, 3, and 4 and rituximab 375 mg/m^2 IV on Day 14, followed by 14 days of rest. Cycles 7-10 (2-month cycle): Following 2 months rest after the completion of Cycle 6, participants with CR, CRu, or PR, received maintenance therapy with rituximab 375 mg/m^2 IV on Day 1, followed by 2 months rest; cycle was repeated 4 times.
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Remaining Failure-Free After 2 Years From Treatment Start Date
Description: Percentage of participants who at 2 years from the start of treatment remained free from documented disease progression, relapse, or death. Failure status was based on tumor evaluation performed on Month 28. Participants who did not have a tumor evaluation at Month 28 were counted as failures.
Time Frame: Month 28
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 46
percentage of participants | 73.9 [61.22 to 86.60]
Statistical Analysis 1: Comparison: Rituximab + Fludarabine + Cyclophosphamide; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

2. Secondary Outcome: Percentage of Participants Achieving a Best Overall Response of CR, CRu, or PR by Study Phase
Description: CR: complete disappearance of all symptoms/objective signs of disease (enlarged lymph nodes, hepatomegaly, splenomegaly) for at least 3 months following definitive re-evaluation at end of therapy. For initial bone marrow involvement, clearance of bone marrow documented by biopsy, normalization of blood counts with granulocytes greater than (>)1,500 per microliter (/µL), hemoglobin >12 grams per deciliter (g/dL), platelets >100,000/µL. CRu: disappearance of all symptoms and nearly all measurable lesions, but persistence of some radiologic abnormalities with normalization of all biologic abnormalities; normalization of the performance status for at least 3 months after the definite evaluation of therapy. PR: at least 50 percent (%) reduction of measurable and evaluable lymphoma involvement for at least 4 weeks without occurrence of new manifestations, normalization of blood counts. Participants without evaluation at end of induction/maintenance phase were considered nonresponders.
Time Frame: Baseline, Months 4, 7 (Induction Phase), 11, 16 (Maintenance Phase),22, 28, 34, and 40(Follow-Up Phase)
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 46
percentage of participants
  Induction Phase | 95.7 [89.76 to 100.00]
  Maintenance Phase | 80.4 [68.97 to 91.90]

3. Secondary Outcome: Percentage of Participants Achieving a Response by Response Type and Study Phase
Description: as for outcome 2
Time Frame: Baseline, Months 4, 7, 11, 16, 22, 28, 34, and 40
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 46
percentage of participants
  CR at end of induction phase | 41.3
  CR at end of maintenance phase | 45.7
  CR at final assessment | 45.7
  CRu at end of induction phase | 21.7
  CRu at end of maintenance phase | 15.2
  CRu at final assessment | 19.6
  PR at end of induction phase | 32.6
  PR at end of maintenance phase | 19.6
  PR at final assessment | 13.0
  Relapse at end of induction phase | 0
  Relapse at end of maintenance phase | 0
  Relapse at final assessment | 2.2
  Unknown at end of induction phase | 4.3
  Unknown at end of maintenance phase | 19.6
  Unknown at final assessment | 19.6

4. Secondary Outcome: Failure-Free Survival (FFS), Percentage of Participants Estimated to be Free of Documented Disease Progression, Relapse, or Death
Description: FFS data were analyzed using Kaplan-Meier survival analysis. FFS was measured from the date of treatment start to the date of documented disease progression, relapse, or death from any cause. Responding participants, participants who were lost to follow up, who withdrew consent, or dropped out due to adverse events (AE) were censored at their last assessment date. The reported data refer to values up to 40 months.
Time Frame: Baseline, Months 1-8, 10-12, 14, 16, 22, 28, 34 and 40
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 46
percentage of participants | 90.12 [75.48 to 96.23]

5. Secondary Outcome: FFS - Percentage of Participants With an Event
Description: FFS was measured from the date of treatment start to the date of documented disease progression, relapse, or death from any cause. Responding participants, participants who were lost to follow up, who withdrew consent, or who dropped out due to AEs were censored at their last assessment date.
Time Frame: Baseline, Months 1-8, 10-12, 14, 16, 22, 28, 34 and 40
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 46
percentage of participants | 8.7

6. Secondary Outcome: FFS - Time to Event
Description: FFS was measured from the date of treatment start to the date of documented disease progression, relapse or death from any cause. Responding participants, participants who were lost to follow up, who withdrew consent or dropped out due to AEs were censored at their last assessment date. NOTE: The mean survival time and its standard error were underestimated because the largest observation was censored and the estimation was restricted to the largest event time.
Time Frame: Baseline, Months 1-8, 10-12, 14, 16, 22, 28, 34 and 40
Population: ITT population
Measure: Mean (Standard Error); unit: months
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 46
months | 39.14 (0.70)

7. Secondary Outcome: Overall Survival (OS) - Percentage of Participants Estimated to be Alive
Description: OS data were analyzed using Kaplan-Meier survival analysis. OS was defined as the time from first dosage of study drug to the date of death from any cause. Reported data refer to values up to 40 months.
Time Frame: Baseline, Months 1-8, 10-12, 14, 16, 22, 28, 34 and 40
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 46
percentage of participants | 97.44 [83.16 to 99.64]

8. Secondary Outcome: OS - Percentage of Participants With an Event
Description: OS was defined as the time from first dosage of study drug to the date of death from any cause.
Time Frame: Baseline, Months 1-8, 10-12, 14, 16, 22, 28, 34 and 40.
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 46
percentage of participants | 2.17

9. Secondary Outcome: OS - Time to Event
Description: Overall survival was defined as the time from first dosage of study drug to the date of death from any cause.
Time Frame: Baseline, Months 1-8, 10-12, 14, 16, 22, 28, 34 and 40.
Population: ITT population
Measure: Mean (Standard Error); unit: months
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 46
months | 38.6 (NA) — Standard error could not be determined because the largest observation was censored and the estimation was restricted to the largest event time.

10. Secondary Outcome: Disease-Free Survival (DFS) - Percentage of Participants Estimated to be Disease-Free
Description: DFS data were analyzed using Kaplan-Meier survival analysis. DFS was defined for all participants who achieved a complete response (CR/CRu) at month 1 after the completion of treatment of the induction phase (Month 7 of the study) and was measured from the time of CR to the date of relapse. Participants without relapse were censored at their last assessment date. Participants who died due to tumour burden were considered in relapse. Participants who died due to any other causes were censored as of the death date. The reported data refer to values up to 40 months.
Time Frame: Baseline, Months 1-8, 10-12, 14, 16, 22, 28, 34 and 40
Population: ITT population; only participants who achieved a complete response (CR/CRu) at month 1 after the completion of treatment of the induction phase were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 29
percentage of participants | 87.70 [65.84 to 95.96]

11. Secondary Outcome: DFS - Percentage of Participants With an Event
Description: DFS was defined for all patients who achieved a complete response (CR/CRu) at month 1 after the completion of treatment of the induction phase (month 7 of the study) and was measured from the time of complete response to the date of relapse. Participants without relapse were censored at their last assessment date. Participants who died due to tumour burden were considered in relapse. Participants who died due to any other causes were censored on the death date.
Time Frame: Baseline, Months 1-8, 10-12, 14, 16, 22, 28, 34 and 40.
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 29
percentage of participants | 10.34

12. Secondary Outcome: DFS - Time to Event
Description: DFS was defined for all participants who achieved a complete response (CR/CRu) at month 1 after the completion of treatment of the induction phase (month 7 of the study) and was measured from the time of complete response to the date of relapse. Participants without relapse were censored at their last assessment date. Participants who died due to tumour burden were considered in relapse. Participants who died due to any other causes were censored on the death date. NOTE: The mean survival time and its standard error were underestimated because the largest observation was censored and the estimation was restricted to the largest event time.
Time Frame: Baseline, Months 1-8, 10-12, 14, 16, 22, 28, 34 and 40.
Population: as for outcome 10
Measure: Mean (Standard Error); unit: months
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 29
months | 32.51 (0.58)

13. Secondary Outcome: Progression-free Survival (PFS) - Percentage of Participants Estimated to Be Progress Free
Description: PFS data were analyzed using Kaplan-Meier survival analysis. PFS was defined as the time from treatment start to the date of documented disease progression. Reported data refer to values up to 40 months.
Time Frame: Baseline, Months 1-8, 10-12, 14, 16, 22, 28, 34 and 40
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 46
percentage of participants | 90.12 [75.48 to 96.23]

14. Secondary Outcome: PFS - Percentage of Participants With an Event
Description: Progression-free survival was defined as the time from the date of treatment start to the date of documented disease progression.
Time Frame: Baseline, Months 1-8, 10-12, 14, 16, 22, 28, 34 and 40
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 46
percentage of participants | 8.70

15. Secondary Outcome: PFS - Time to Event
Description: Progression-free survival was defined as the time from treatment start to the date of documented disease progression. NOTE: The mean survival time and its standard error were underestimated because the largest observation was censored and the estimation was restricted to the largest event time.
Time Frame: Baseline, Months 1-8, 10-12, 14, 16, 22, 28, 34 and 40
Population: ITT population
Measure: Mean (Standard Error); unit: months
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 46
months | 39.14 (0.70)

16. Secondary Outcome: Duration of Response (DR) - Percentage of Participants Expected to Maintain a Response
Description: DR data were analyzed using Kaplan-Meier survival analysis. DR was defined for all participants who achieved a response (CR, CRu and PR) at month 1 after the completion of treatment of the induction phase (Month 7 of the study) and was measured from the time of response until the date of progression or relapse. Participants without relapse or progression were censored at their last assessment date. Participants who died due to tumour were considered in progression. Participants who died for any other cause were censored to the death date.
Time Frame: Baseline, Months 1-8, 10-12, 14, 16, 22, 28, 34 and 40
Population: ITT population; only participants who achieved a response (CR, CRu and PR) at month 1 after the completion of treatment of the induction phase of the study were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 44
percentage of participants | 90.07 [75.45 to 96.19]

17. Secondary Outcome: DR - Percentage of Participants With an Event
Description: DR was defined for all participants who achieved a response (CR, CRu and PR) at month 1 after the completion of treatment of the induction phase (Month 7 of the study) and was measured from the time of response until the date of progression or relapse. Participants without relapse or progression were censored at their last assessment date. Participants who died due to tumour were considered in progression. Participants who died for any other cause were censored to the death date.
Time Frame: Baseline, Months 1-8, 10-12, 14, 16, 22, 28, 34 and 40
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 44
percentage of participants | 9.09

18. Secondary Outcome: DR - Time to Event
Description: as for outcome 17
Time Frame: Baseline, Months 1-8, 10-12, 14, 16, 22, 28, 34 and 40
Population: ITT population: only participants who achieved a response (CR, CRu and PR) at month 1 after the completion of treatment of the induction phase of the study were included in the analysis.
Measure: Mean (Standard Error); unit: months
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 44
months | 32.19 (0.72)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (AEs) were reported throughout the study (up to 40 months).
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Serious Adverse Events (participants affected / at risk) | 16/47
Other Adverse Events (participants affected / at risk) | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Fludarabine + Cyclophosphamide (N=47)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Mitral valve incompetence (Cardiac disorders) | 1
Renal dysplasia (Congenital, familial and genetic disorders) | 1
Pyrexia (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Bronchopneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Staphylococcal infection (Infections and infestations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Fludarabine + Cyclophosphamide (N=47)
Anaemia (Blood and lymphatic system disorders) | 8
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 18
Neutropenia (Blood and lymphatic system disorders) | 29
Pancytopenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Hydrocele (Congenital, familial and genetic disorders) | 2
Ear pain (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Conjunctivitis (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Visual disturbance (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 5
Dysphagia (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 20
Stomatitis (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 5
Asthenia (General disorders) | 16
Chills (General disorders) | 2
Fatigue (General disorders) | 1
Hyperthermia (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 2
Pain (General disorders) | 4
Pyrexia (General disorders) | 23
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Allergy to arthropod bite (Immune system disorders) | 1
Amyloidosis (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Hypogammaglobulinaemia (Immune system disorders) | 5
Bronchitis (Infections and infestations) | 6
Conjunctivitis infective (Infections and infestations) | 1
Conjunctivitis viral (Infections and infestations) | 1
Cystitis (Infections and infestations) | 2
Ear infection (Infections and infestations) | 2
Erythema induratum (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Haemophilus infection (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 8
Influenza (Infections and infestations) | 2
Labyrinthitis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Pulmonary mycosis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Beta 2 microglobulin increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 2
Red blood cell sedimentation rate increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Amnesia (Nervous system disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Neuropathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 2
Polyuria (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Renal pain (Renal and urinary disorders) | 1
Amenorrhoea (Reproductive system and breast disorders) | 1
Gynaecomasatia (Reproductive system and breast disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 2
Periorbital oedema (Skin and subcutaneous tissue disorders) | 1
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 4
Skin fissures (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Ureterectomy (Surgical and medical procedures) | 1
Aortic thrombosis (Vascular disorders) | 1
Flushing (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 1
Raynaud's phenomenon (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request the Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.